CLINICAL TRIAL: NCT00005993
Title: Immunotherapy With Subcutaneous Il-2 and Stem Cell Factor (SCF) for Patients With Lymphoma or Breast Cancer After Autologous Transplantation
Brief Title: Biological Therapies Following Peripheral Stem Cell Transplantation in Treating Patients With Non-Hodgkin's Lymphoma, Hodgkin's Disease, or Advanced Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 1999LS022; MT1998-21 (Other: Blood and Marrow Transplantation Program); NCI-G00-1803
Record Dates: First submitted 2000-07-05; First posted 2004-06-21 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Breast Cancer; Lymphoma
Keywords: stage IV breast cancer; stage IIIA breast cancer; recurrent breast cancer; stage IIIB breast cancer; recurrent adult Hodgkin lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Breast Neoplasms; Lymphoma; Hodgkin Disease; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — aldesleukin; Filgrastim; Stem Cell Factor; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: aldesleukin
Drug: filgrastim
Drug: recombinant human stem cell factor
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Interleukin-2 may stimulate a person's white blood cells to kill cancer cells. Filgrastim and stem cell factor may increase the number of immune cells found in bone marrow or peripheral blood and may help a person's immune system recover from the side effects of cancer therapy. Peripheral stem cell transplantation may be able to replace immune cells that were destroyed by therapy used to kill cancer cells.

PURPOSE: Phase I trial to study the effectiveness of interleukin-2 and stem cell factor following peripheral stem cell transplantation in treating patients who have non-Hodgkin's lymphoma, Hodgkin's disease, or advanced breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety and maximum tolerated dose of interleukin-2 (IL-2) and stem cell factor (SCF) following autologous peripheral blood stem cell transplantation in patients with non-Hodgkin's lymphoma or advanced breast cancer. II. Determine the effectiveness of filgrastim (G-CSF) and SCF as mobilizing agents in these patients.

OUTLINE: This is a dose escalation study of stem cell factor (SCF). Patients receive filgrastim (G-CSF) subcutaneously (SC) followed by SCF SC daily for 7-10 days. Beginning on the fifth day of G-CSF and SCF injections, peripheral blood stem cells (PBSC) are collected over several days. PBSC are later reinfused and patients receive G-CSF SC daily until hematopoietic recovery. At least 30 days but no later than 110 days following transplant, patients who did not experience adverse reactions to SCF during mobilization begin posttransplant immunotherapy. Patients receive interleukin-2 SC daily and SCF SC 3 times weekly for 6 weeks. Treatment continues in the absence of unacceptable toxicity or disease progression. Cohorts of 3-6 patients receive escalating doses of SCF during posttransplant immunotherapy until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose limiting toxicities. Patients are followed at 1 week, every 3 months for 1 year, and then every 6 months thereafter.

PROJECTED ACCRUAL: A maximum of 27 patients will be accrued for this study within 1-1.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Hodgkin's disease, non-Hodgkin's lymphoma, or advanced stage breast cancer Planned treatment is autologous peripheral blood stem cell transplantation No T-cell lymphomas Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 18 to 65 Menopausal status: Not specified Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Immunologic: No history of seasonal or recurrent asthma within the past 5 years No concurrent asthmatic symptoms (e.g., wheezing) related to a current respiratory tract infection No anaphylactic/anaphylactoid type event manifested by disseminated urticaria, laryngeal edema, hypotension, and/or bronchospasm (e.g., food or insect venom) within the past 5 years Drug allergies manifested solely by rash allowed No history of angioedema or recurrent urticaria lasting longer than 14 days No history of hereditary or acquired angioedema No known allergy to E. coli derived products Other: Not pregnant Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics At least 1 week since prior hematopoietic growth factors Chemotherapy: Not specified Endocrine therapy: No concurrent steroids Radiotherapy: No concurrent radiotherapy Surgery: Not specified Other: No concurrent beta adrenergic blocking agents No concurrent therapeutic antibiotics posttransplant No concurrent IV hyperalimentation or IV fluids posttransplant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-05; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda J. Burns, MD, Study Chair — Masonic Cancer Center, University of Minnesota